CLINICAL TRIAL: NCT03828253
Title: Ellipsys Percutaneous Arteriovenous Fistula for Hemodialysis Access
Brief Title: Ellipsys Fistula for Hemodialysis Access
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Richmond Vascular Center (Other)
Responsible Party: Sponsor
Other Study IDs: pAVF 1.0
Record Dates: First submitted 2018-10-18; First posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To report the outcomes of patients having percutaneous proximal radial artery fistula creation.

DETAILED DESCRIPTION:
The study would like to enroll up to 100 patients without age, gender-based, race and ethnicity enrollment restrictions for adults over 18 years of age. Women of child bearing potential are not excluded. If a pregnant patient required, an arteriovenous fistula for hemodialysis an Ellipsys® fistula would be an option. The Investigator would like to consent previous Ellipsys® patients with appropriate medical records so that the Investigator may capture participants data for outcomes reporting.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18 years or older
* Diagnosed with ESRD or chronic kidney disease requiring dialysis or anticipating start of dialysis
* Adjacent vein diameter of > 2.0 mm at target anastomosis site and confirmed clinically significant outflow
* Arterial lumen diameter of > 2.0 mm at target anastomosis site
* Adequate collateral arterial perfusion: Barbeau test grade A through C
* Radial artery -adjacent vein proximity < 1.5 mm measured lumen edge-to-lumen edge via ultrasound

Exclusion Criteria:

* Target vessel that are < 2mm is diameter
* Distance between the target artery and vein > 1.5 mm
* Edema of the upper extremity on the ipsilateral side
* Barbeau test grade D

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Recruitment of subjects will be from the current End Stage Renal disease patient population at Richmond Vascular Center and referrals from Nephrologists and Vascular Surgeons.
  The study would like to enroll up to 100 patients without age, gender-based, race and ethnicity enrollment restrictions for adults over 18 years of age. Women of child bearing potential are not excluded. If a pregnant patient required, an arteriovenous fistula for hemodialysis an Ellipsys® fistula would be an option. We would like to consent previous Ellipsys® patients with appropriate medical records so that we may capture their data for outcomes reporting.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-08-27 (Estimated); Study Completion 2021-08-27 (Estimated)

PRIMARY OUTCOMES:
Blood flow Volume | 90 days
  Brachial Artery flow volume of 500ml as measured on Ultrasound Duplex

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Hull, MD, Principal Investigator — Richmond Vascular Center
Locations (1):
- Richmond Vascular Center, North Chesterfield, Virginia, United States

REFERENCES:
- [Derived] Hull J, Deitrick J, Groome K. Maturation for Hemodialysis in the Ellipsys Post-Market Registry. J Vasc Interv Radiol. 2020 Sep;31(9):1373-1381. doi: 10.1016/j.jvir.2020.03.001. Epub 2020 Aug 14. PMID 32800660